CLINICAL TRIAL: NCT03470896
Title: Quality of Preanesthesia Teleconsultation Versus Preanesthesia Traditional Consultation : a Randomized Controlled Equivalence Trial.
Brief Title: Quality of Preanesthesia Teleconsultation : a Randomized Controlled Trial.
Acronym: TELECAM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2017-A03084-49
Record Dates: First submitted 2018-03-08; First posted 2018-03-20 (Actual); Last update posted 2018-03-20 (Actual); Status verified 2018-01

CONDITIONS: Preanesthesia Consultation
Keywords: preanesthesia teleconsultation; video-conference; ambulatory surgery; telemedicine

STUDY DESIGN:
Intervention Model Description: One group : preanesthesia teleconsultation / One group : preanesthesia traditional teleconsultation / One sub-group : bis preanesthesia traditional teleconsultation
Who Masked: Outcomes Assessor
Masking Description: Participant and care provider know the allocation group "teleconsultation" or "traditional consultation".
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Preanesthesia teleconsultation (Active Comparator): Preanesthesia teleconsultation through video-conference, between an anesthesiologist of the surgical center Emile Galle, in a medical consulting room in the surgical center Emile Galle, and a patient at home or at work. The patient must be in a quiet area, which allows the confidential medical contact.
  Interventions: Procedure: preanesthesia teleconsultation
- Preanesthesia traditional consultation (Active Comparator): Preanesthesia traditional consultation between an anesthesiologist of the surgical center Emile Galle, and a patient, in a medical consulting room in the surgical center Emile Galle.
  Interventions: Procedure: preanesthesia traditional consultation
- Bis traditional consultation (Other): If a patient, in the group " preanesthesia teleconsultation " cannot realized his teleconsultation because of technical problem, he will be assigned on the sub group " bis traditional preanesthesia consultation ".
  Interventions: Procedure: preanesthesia traditional consultation

INTERVENTIONS:
Procedure: preanesthesia teleconsultation — According to his allocated group, patient will have a teleconsultation at home/at work with an anaesthesiologist.
  Arms: Preanesthesia teleconsultation
Procedure: preanesthesia traditional consultation — According to his allocated group, patient will have a traditional consultation with an anaesthesiologist in the surgical center Emile Galle.
  Arms: Bis traditional consultation; Preanesthesia traditional consultation

SUMMARY:
Since the publication of the law " Hôpital, Patients, Santé, Territoire " of 2009 in France, the development of telemedicine is a public health issue. It is also a government priority registered in the government investment plan of 2017-2018.

The quality of preanesthesia teleconsultation at home, through video-conference, has never been tested in practice.The aim of this study is to evaluate the quality of preanesthesia teleconsultations through video-conference, compared with traditional preanesthesia consultations. The quality is established by the assessment of the primary outcome : the risks related to difficult intubation, in patients undergoing ambulatory surgery at the Surgical Center Emile Galle. Our research hypothesis is that there is no difference between the quality of preanesthesia teleconsultations through video-conference, and the quality of traditional preanesthesia consultations. Secondary objectives are to identify satisfaction and preoperative anxiety of patients regarding teleconsultation, to identify satisfaction of practioners regarding teleconsultation, to evaluate the quality (based on the assessment of secondary outcomes) of preanesthesia teleconsultations compared with traditional preanesthesia consultations, and to evaluate the technical viability of generalising preanesthesia teleconsultation.

ELIGIBILITY:
Inclusion Criteria:

* Patient with social security affiliation.
* Informed consent from patient
* Patient with an ambulatory surgery programmed in the surgical center Emile Galle (CHRU de Nancy)
* Patient with technology equipments, which are compatible with the plateform of video-conference :
* smartphones, touch pads, computer
* web-browser ( chrome or internet explorer)
* Webcam and microphone
* Printer

Exclusion Criteria:

* Patients covered by Articles L. 1121-5 to L. 1121-8, L1122-2 and L. 1122-1-2 of the french public health code. (Persons especially protected by Act)
* Patients refusing to participate to the study, or refusing the randomization for the group allocation.
* Preanesthesia consultation for a programmed surgery in an hospital other than the surgical center of Emile Galle.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2018-05-01 (Estimated); Primary Completion 2021-05 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
Agreement concerning the risk of difficult intubation between preanesthesia consultation and visit. | 1 day before surgery or baseline (J0 = surgery day)
  The quality of a preanesthesia consultation (teleconsultations or traditional consultations) is considered to be correct when the result (presence or lack of difficult intubation risks) is consistent with the result of the preanesthesia visit (before surgery.) If yes from 2 of the 4 following propositions about predictable intubation difficulty ( mallampi score > II (yes/no), previous difficult intubation (yes/no), oral opening <30mm (yes/no), distance thyro-mentonnière < 65mm. (yes/no)), the predictable intubation will be difficult.

SECONDARY OUTCOMES:
Agreement between preanesthesia consultation and visit concerning the risk of difficult mask ventilation | 1 day before surgery or baseline (J0 = surgery day)
  The quality of a preanesthesia consultation (teleconsultations or traditional consultations) is considered to be correct when the result (presence or lack of difficult mask ventilation risks) is consistent with the result of the preanesthesia visit (before surgery.) If yes from 2 of the 4 following propositions about predictable mask ventilation difficulty ( patient with a barbe (yes/no), BMI>26 kg/m2 (yes/no), edentulous patient (yes/no), an age > 55 years old (yes/no)), snoring (yes/no), the predictable mask ventilation will be difficult.
Agreement between preanesthesia consultation and visit concerning the evaluation of "American Society of Anesthesiologists" (ASA) score of the patient | 1 day before surgery or baseline (J0 = surgery day)
  The quality of a preanesthesia consultation (teleconsultations or traditional consultations) is considered to be correct when the result (ASA score of the patient) is consistent with the result of the preanesthesia visit (before surgery.)
Agreement between preanesthesia consultation and visit concerning correct treatment management. | 1 day before surgery or baseline (J0 = surgery day)
  The quality of a preanesthesia consultation (teleconsultations or traditional consultations) is considered to be correct when the result (treatment management : interruption, continuation, relay) is consistent with the result of the preanesthesia visit (before surgery.)
Agreement between preanesthesia consultation and visit concerning completeness of preoperative workup | 1 day before surgery or baseline (J0 = surgery day)
  The quality of a preanesthesia consultation (teleconsultations or traditional consultations) is considered to be correct when the result (preoperative workup : complete blood count (CBC) with platelet or/and coagulation factors or/and ionograms or/and blood group, or/and consultation with a specialist physician ) is consistent with the result of the preanesthesia visit (before surgery.)
Satisfaction of anesthesiologist | 1 day before surgery or baseline (J0 = surgery day)
  Satisfaction of anesthesiologist, who realized teleconsultation, tested by visual analogue scale : from 0 to 10 (poor to good results), in comparison with traditional consultation
Satisfaction of patient | 1 day before surgery or baseline (J0 = surgery day)
  Satisfaction of patient, who attended teleconsultation, tested by visual analogue scale : from 0 to 10 (poor to good results) in comparison with traditional consultation
Preoperative anxiety of patient | 1 day before surgery or baseline (J0 = surgery day)
  Preoperative anxiety of patient, who attended teleconsultation, tested by amsterdam scale (APAIS), in comparison with traditional consultation
Calculation of a ratio to evaluate the technical viability of generalising preanesthesia teleconsultation | 1 day before surgery or baseline (J0 = surgery day)
  evaluate the technical viability of generalising preanesthesia teleconsultation, with calculation of ratio : number of randomized patients in group " preanesthesia teleconsultation ", who finally get a teleconsultation / number of randomized patients in group " preanesthesia teleconsultation. " The higher the ratio, the higher the teleconsultation can be considered as a generalisable care practice.

CONTACTS AND LOCATIONS:
Overall Officials: Herve BOUAZIZ, PUPH, Principal Investigator — Central HNF

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Roche A, Simon M, Bouaziz H, Poussel M, Sirveaux F, Adam I, Delpuech M, Thilly N. Quality of Preanesthesia Teleconsultation: The TELECAM Randomized Controlled Trial. Telemed J E Health. 2024 Aug;30(8):e2300-e2310. doi: 10.1089/tmj.2024.0027. Epub 2024 May 3. PMID 38700568